CLINICAL TRIAL: NCT02103218
Title: A Risky Sex Prevention Intervention for Middle School Age Minority Girls
Acronym: GEMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Greensboro (Other)
Responsible Party: Principal Investigator, Dr. Tracy R. Bartlett, Associate Professor, University of North Carolina, Greensboro
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P20MD002289-1; P20MD002289 (NIH)
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-05

CONDITIONS: HIV; Risky Sex Prevention
Keywords: HIV; risky sex prevention; intervention
MeSH Terms: interventions — Educational Status; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risky sex prevention (Experimental): education, activities, empowerment, racial pride building
  Interventions: Behavioral: Education, activities, empowerment, racial pride building
- Healthy behaviors (Active Comparator): General health education, activities
  Interventions: Behavioral: General Health education, activities

INTERVENTIONS:
Behavioral: Education, activities, empowerment, racial pride building — Intervention focuses on information aimed toward reducing or preventing risky sex behaviors of minority adolescent females.
  Arms: Risky sex prevention
Behavioral: General Health education, activities — Intervention focuses on information regarding general health knowledge and healthy behaviors (not including sex).
  Arms: Healthy behaviors

SUMMARY:
African American adolescent females are more likely to have sex at an early age, to have older sex partners that have had multiple sexual experiences, and are less likely to use a condom than their white counterparts. Lack of sexual assertiveness is a factor in the risky sex behaviors of young African American women. African American girls at the greatest risk for contracting HIV are the ones that report that their partners could convince them to have sex and report trouble communicating their wishes related to sex. Thus far no intervention has addressed the disparate rate of HIV infection in young African American girls. This study is unique in promoting increases in racial pride as a component of empowerment to help African American girls self-protect against HIV. The study has the potential to empower young African American girls to delay sex initiation or reduce risky sex behaviors and thus reduce their risk of contracting HIV.

DETAILED DESCRIPTION:
This is a longitudinal intervention study with a study condition intervention and a control condition intervention. Potential participants will be invited to a recruitment meeting. If they choose to participate, they will be asked to sign informed consent or assent. There are 4 data collections for moms and girls - 1 after recruitment but before the start of the intervention, 1 at the end of the intervention (after the girls 12 week intervention), 1 three months after the end of the intervention (about 6 months after recruitment), and the final data collection 9 months after the end of the intervention (about 12 months from recruitment). Girls are asked to attend 12 group intervention sessions of about 2 hours each, once weekly, and then a final termination session that is followed by a celebration session to which their mothers are invited and then an evaluation session. Moms are asked to participate in 3 one hour education sessions over the 12 weeks that their daughters are in the weekly sessions, the celebration with their daughters, and then their evaluation session. Moms will also be asked to give their daughter empowering messages 5-7 times/week and girls asked to receive them. Finally, moms will be asked to receive calls from the study team once per month or 1 year to be asked about the empowering messages they have been sending their daughters.

ELIGIBILITY:
Mother Inclusion Criteria:

* Must be 21 years or older.
* Must be daughter's primary female guardian/caregiver and she lives with me at least 50% of the time.
* Must understand spoken and written English.
* Must be able to provide a phone number where they can be reached and will be able to maintain contact with researchers for one year after start of study.
* Must be able to provide or arrange reliable transportation for their daughter after each session or data collection.

Mother Exclusion Criteria:

* Must not be incarcerated at the time of recruitment
* Must not have a physical or mental health condition that may affect my or my daughter's participation in the study.

Daughter Inclusion Criteria:

* Must be in middle school (grades 6-8) at the time of recruitment.
* Must be between the ages of 11-14 at the time of recruitment.
* Must self-identify as Black, African-American, or a mixed race that includes black or African-American.
* Must be able to understand written and spoken English.

Daughter Exclusion Criteria:

* Must not be in a classroom for developmentally delayed students in school.
* Must not be currently pregnant at the time of recruitment.
* Must not have a mental or physical health condition that may affect her participation in the study.
* Must not be suspended or expelled from school at the time of recruitment.

Ages: 11 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2012-11; Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy R Bartlett, PhD, Principal Investigator — University of North Carolina, Greensboro; Debra C Wallace, PhD, Study Chair — Univeristy of North Carolina, Greensboro
Locations (1):
- University of North Carolina, Greensboro, Greensboro, North Carolina, United States

REFERENCES:
- [Background] Wallace DC, Bartlett R. Recruitment and retention of African American and Hispanic girls and women in research. Public Health Nurs. 2013 Mar;30(2):159-66. doi: 10.1111/phn.12014. Epub 2012 Nov 22. PMID 23452110
- [Result] Bartlett R, Johnson A, Randolph I, McCoy TP. Communication and Bonding Between African-American Middle School Girls and Their Maternal Figures. J Natl Black Nurses Assoc. 2016 Jul;27(1):18-23. PMID 29932539

RESULTS

PARTICIPANT FLOW:
Groups:
- Risky Sex Prevention-Daughters: Education, activities, empowerment, racial pride building...
- Healthy Behaviors-Daughters; Healthy Behaviors-Mothers: General health education, activities
- Risky Sex Prevention-Mothers: Activities, empowerment, communication...
Period: Overall Study
Arm/Group | Risky Sex Prevention-Daughters | Healthy Behaviors-Daughters | Risky Sex Prevention-Mothers | Healthy Behaviors-Mothers
Started | 51 | 59 | 48 | 54
Completed | 46 | 51 | 44 | 47
Not Completed | 5 | 8 | 4 | 7

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants (212) is based on both daughters and mothers in all arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Risky Sex Prevention-Daughters | Healthy Behaviors-Daughters | Risky Sex Prevention-Mothers | Healthy Behaviors-Mothers | Total
Number analyzed (Participants) | 51 | 59 | 48 | 54 | 212
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (0.70) | 12.7 (0.94) | 40.9 (10.3) | 37.8 (6.39) | 25.7 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 59 | 48 | 54 | 212
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: African-American | 30 | 48 | 38 | 48 | 164
  Race/Ethnicity: Mixed | 21 | 11 | 6 | 2 | 40
  Race/Ethnicity: Hispanic/Latino | 0 | 0 | 2 | 0 | 2
  Race/Ethnicity: Other | 0 | 0 | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 51 | 59 | 48 | 54 | 212
Current Grade [Count of Participants; unit: Participants] — Population: Only daughters (n=110) were analyzed for middle school grade.
  Participants
    number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    6th grade | 22 | 21 |  |  | 43
    7th grade | 23 | 21 |  |  | 44
    8th grade | 6 | 17 |  |  | 23
Racial Pride [Mean (Standard Deviation); unit: units on a scale] — Population: This measure was not assessed for Mothers.
  units on a scale
    number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    (all) | 21.0 (4.2) | 21.3 (4.3) |  |  | 21.2 (4.3)
Maternal Monitoring Scale [Mean (Standard Deviation); unit: units on a scale] — There are two separate scales: One asked from the perspective of the daughter and one asked from the perspective of the mother. They should be kept separate as has previous literature. For example, they each have their own estimated scale reliability (alpha = .70 for daughters and alpha = .58 for mothers) and should NOT be averaged over daughters and mothers. Population: Two separate scales: From daughter's perspective and mother's perspective. Should be kept separate like previous literature. They each have their own reliability (alpha = .70 for daughters and .58 for mothers) and should NOT be averaged over daughters and mothers. We therefore present data by 2 rows: (a) for Daughters only and (b) for Mothers only.
  units on a scale
    Daughters only: number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    Daughters only | 34.8 (4.2) | 35.2 (4.3) |  |  | 35.0 (4.2)
    Mothers only: number analyzed (Participants) | 0 | 0 | 48 | 54 | 102
    Mothers only |  |  | 37.4 (2.6) | 37.4 (2.2) | 37.4 (2.4)
Mother-Adolescent Communication: Open Family Communication [Mean (Standard Deviation); unit: units on a scale] — There are two separate scales: One asked from the perspective of the daughter and one asked from the perspective of the mother. They should be kept separate as has previous literature. For example, they each have their own estimated scale reliability (alpha = .87 for daughters and alpha = .70 for mothers) and should NOT be averaged over daughters and mothers. We therefore reported as separate rows for Daughters only and Mothers only. Population: Two separate scales: One from daughter's perspective and mother's perspective. They should be kept separate like previous literature. They each have their own reliability (alpha = .87 for daughters and alpha = .70 for mothers) and should NOT be averaged over daughters and mothers. We therefore reported as separate by Daughters and Mothers.
  units on a scale
    Daughters only: number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    Daughters only | 38.1 (9.0) | 40.6 (7.7) |  |  | 39.4 (8.4)
    Mothers only: number analyzed (Participants) | 0 | 0 | 48 | 54 | 102
    Mothers only |  |  | 41.1 (5.2) | 41.2 (5.3) | 41.1 (5.3)
Mother-Teen Sexual Risk Communication [Mean (Standard Deviation); unit: units on a scale] — Population: This measure was only collected for daughters (n=110).
  units on a scale
    number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    (all) | 24.5 (8.6) | 24.2 (9.1) |  |  | 24.4 (8.8)
HIV Knowledge [Mean (Standard Deviation); unit: units on a scale] — Population: This measure was only collected for daughters (n=110).
  units on a scale
    number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    (all) | 9.9 (2.5) | 9.1 (3.2) |  |  | 9.5 (2.9)
Maternal Bond Scale [Mean (Standard Deviation); unit: units on a scale] — Population: This measure was only collected for daughters (n=110).
  units on a scale
    number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    (all) | 26.3 (5.9) | 27.9 (4.5) |  |  | 27.2 (5.2)
Rosenberg Self-Esteem [Mean (Standard Deviation); unit: units on a scale] — Population: This measure was only collected for daughters (n=110).
  units on a scale
    number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    (all) | 21.0 (5.9) | 21.8 (4.2) |  |  | 21.5 (5.0)
Sexual Assertiveness: Refusal subscale [Mean (Standard Deviation); unit: units on a scale] — Population: This measure was only collected for daughters (n=110).
  units on a scale
    number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    (all) | 23.3 (5.2) | 23.9 (4.9) |  |  | 23.6 (5.0)
Sexual Assertiveness: Prevent subscale [Mean (Standard Deviation); unit: units on a scale] — Population: This measure was only collected for daughters (n=110).
  units on a scale
    number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    (all) | 27.0 (4.3) | 25.5 (4.9) |  |  | 26.2 (4.7)
Empowerment: Interpersonal [Mean (Standard Deviation); unit: units on a scale] — Population: This measure was only collected for daughters (n=110).
  units on a scale
    number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    (all) | 9.4 (2.2) | 9.2 (2.6) |  |  | 9.3 (2.4)
Empowerment: Relationship [Mean (Standard Deviation); unit: units on a scale] — Population: This measure was only collected for daughters (n=110).
  units on a scale
    number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    (all) | 8.0 (4.0) | 7.9 (3.8) |  |  | 8.0 (3.9)
Empowerment: Personal [Mean (Standard Deviation); unit: units on a scale] — Population: This measure was only collected for daughters (n=110).
  units on a scale
    number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    (all) | 18.5 (2.6) | 18.2 (4.2) |  |  | 18.4 (3.5)
Adolescent Sexual Activity Index [Mean (Standard Deviation); unit: units on a scale] — Population: This measure was only collected for daughters (n=110).
  units on a scale
    number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    (all) | 1.5 (1.6) | 1.5 (1.6) |  |  | 1.5 (1.7)
Any sex no condom, past 3 months [Count of Participants; unit: Participants] — Population: This measure was only collected for daughters (n=110).
  Participants
    number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    (all) | 4 | 1 |  |  | 5
Sex with multiple partners, ever [Count of Participants; unit: Participants] — Population: This measure was only collected for daughters (n=110).
  Participants
    number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    (all) | 1 | 2 |  |  | 3
Drugs/Alcohol use during sex, past 3 months [Count of Participants; unit: Participants] — Population: This measure was only collected for daughters (n=110).
  Participants
    number analyzed (Participants) | 51 | 59 | 0 | 0 | 110
    (all) | 2 | 0 |  |  | 2
Communication about Sex Self-Efficacy [Mean (Standard Deviation); unit: units on a scale] — 12 items; Cronbach's alpha = .78. Population: This measure was only collected for mothers (n=102).
  units on a scale
    number analyzed (Participants) | 0 | 0 | 48 | 54 | 102
    (all) |  |  | 55.8 (5.3) | 55.8 (5.2) | 55.8 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Adolescent Sexual Activity Index
Description: Adolescent Sexual Activity Index (Female). The theoretical minimum and maximum values are min=0 and max=10 (Hansen, Paskett, & Carter, 1999). A higher index value indicates more activity (worse outcome).
Time Frame: 12 months
Population: Analyses were performed after multiple imputation for missing data. Number at 12 months before imputation were n=46 for Risky sex prevention and n=51 for Health behaviors.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 51 | 59
score on a scale
  Baseline / Pre-Interveniton | 1.39 (.19) | 1.45 (.19)
  At 12 months | 2.12 (.33) | 1.90 (.30)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; Results from count GEE models for outcome with IPW propensity score adjustment and multiple imputation for missing data. Numbers presented above are model-based least-squares means, (SE). Overall p-values from omnibus test (group by time interaction) for any differences in change over time between groups as well as p-values from testing difference in least-square mean estimates in post-hoc pairwise comparisons with pre-intervention were estimated; Test type: Superiority; p = 0.62, count GEE

2. Primary Outcome: Any Sex no Condom, Past 3 Months
Description: Any sex no condom, past 3 months
Time Frame: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: logistic GEE predicted probability as %
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 51 | 59
logistic GEE predicted probability as %
  Baseline / Pre-Interveniton | 7.1 (3.6) | 1.3 (1.3)
  At 12 months | 8.4 (4.3) | 2.4 (1.7)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; Results from logistic GEE models for outcome with IPW propensity score adjustment and multiple imputation for missing data. Numbers presented above are model-based least-squares predicted probabilities converted to %, (SE). Overall p-values from omnibus test (group by time interaction) for any differences in change over time between groups as well as p-values from testing difference in least-square estimates in post-hoc pairwise comparisons with pre-intervention were estimated; Test type: Superiority; p = 0.15, logistic GEE

3. Primary Outcome: Sex With Multiple Partners, Ever
Description: Sex with multiple partners, ever
Time Frame: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: logistic GEE predicted probability as %
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 51 | 59
logistic GEE predicted probability as %
  Baseline / Pre-Interveniton | 0.0 (0.0) | 0.0 (0.0)
  At 12 months | 1.0 (0.9) | 2.2 (1.3)
Statistical Analysis 1: Comparison: Risky Sex Prevention; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.47, logistic GEE

4. Primary Outcome: Drugs/Alcohol Use During Sex, Past 3 Months
Description: Drugs/Alcohol use during sex, past 3 months
Time Frame: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: logistic GEE predicted probability as %
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 51 | 59
logistic GEE predicted probability as %
  Baseline / Pre-Interveniton | 4.4 (3.2) | 0.0 (0.0)
  At 12 months | 1.3 (1.4) | 5.1 (3.7)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.29, logistic GEE

5. Secondary Outcome: HIV Knowledge
Description: HIV-Knowledge Questionnaire for Adolescent Girls. The theoretical minimum and maximum values are min=0 and max=18. Higher scores indicate higher HIV knowledge which is a better outcome.
Time Frame: 12 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 51 | 59
score on a scale
  Baseline / Pre-Interveniton | 9.8 (0.31) | 8.5 (0.56)
  At 12 months | 13.1 (0.38) | 10.4 (0.35)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; Results from linear GEE models for outcome with IPW propensity score adjustment and multiple imputation for missing data. Numbers presented above are model-based least-squares means, (SE). Overall p-values from omnibus test (group by time interaction) for any differences in change over time between groups as well as p-values from testing difference in least-square mean estimates in post-hoc pairwise comparisons with pre-intervention were estimated; Test type: Superiority; p < 0.001, linear GEE

6. Secondary Outcome: Maternal Bond Scale
Description: Maternal Bond Scale. The theoretical minimum and maximum are min=8 to max=40. Higher scores indicate stronger maternal bonds which is a better outcome.
Time Frame: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 51 | 59
score on a scale
  Baseline / Pre-Interveniton | 26.9 (0.78) | 27.8 (0.62)
  At 12 months | 26.8 (0.63) | 28.9 (0.65)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.02, linear GEE — Omnibus overall test for any group x time interaction was p = 0.77

7. Secondary Outcome: Mother-Teen Sexual Risk Communication
Description: Mother-Teen Sexual Risk Communication. The theoretical minimum and maximum are min=8 to max=40. Higher scores indicate greater mother-teen communication about sexual risk which is a better outcome.
Time Frame: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 51 | 59
score on a scale
  Baseline / Pre-Interveniton | 22.8 (1.4) | 22.0 (1.6)
  At 12 months | 25.4 (1.1) | 26.1 (1.4)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.67, linear GEE

8. Secondary Outcome: Mother-Adolescent Communication: Open Family Communication (Girl)
Description: Mother-Adolescent Communication: Open Family Communication (Girl). The theoretical minimum and maximum values are min=10 and max=50. A higher value indicates greater mother-adolescent open family communication which is a better outcome.
Time Frame: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 51 | 59
score on a scale
  Baseline / Pre-Interveniton | 39.1 (1.1) | 39.5 (1.6)
  At 12 months | 37.8 (1.3) | 39.2 (1.2)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.45, count GEE

9. Secondary Outcome: Maternal Monitoring Scale (Girl)
Description: Maternal Monitoring Scale (Girl). The theoretical minimum and maximum values are min=8 and max=40. A higher value indicates greater maternal monitoring which is a better outcome.
Time Frame: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 51 | 59
score on a scale
  Baseline / Pre-Interveniton | 34.4 (0.76) | 35.0 (0.50)
  At 12 months | 34.7 (0.67) | 35.1 (0.78)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.70, count GEE

10. Secondary Outcome: Rosenberg Self-Esteem
Description: Rosenberg Self-Esteem Scale. The theoretical minimum and maximum values are min=10 and max=40. A higher value indicates higher self-esteem which is a better outcome.
Time Frame: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 51 | 59
score on a scale
  Baseline / Pre-Interveniton | 20.6 (0.88) | 21.7 (0.64)
  At 12 months | 21.8 (1.0) | 22.8 (0.90)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.42, linear GEE

11. Secondary Outcome: Racial Pride
Description: Racial Pride Scale. The theoretical minimum and maximum values are min=7 and max=28. A higher value indicates stronger feelings of racial pride which is a better outcome.
Time Frame: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 51 | 59
score on a scale
  Baseline / Pre-Interveniton | 20.9 (0.71) | 21.2 (0.54)
  At 12 months | 22.7 (0.52) | 22.3 (0.56)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.63, count GEE

12. Secondary Outcome: Empowerment: Interpersonal
Description: Empowerment Scale: Interpersonal. The theoretical minimum and maximum values are min=4 and max=20. A higher value indicates greater personal influence on relationship decisions.
Time Frame: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 51 | 59
score on a scale
  Baseline / Pre-Interveniton | 14.7 (0.32) | 14.8 (0.36)
  At 12 months | 14.2 (0.35) | 15.2 (0.30)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.05, count GEE — Omnibus overall test for any group x time interaction was p = 0.78

13. Secondary Outcome: Empowerment: Relationship
Description: Empowerment Scale: Interpersonal. The theoretical minimum and maximum values are min=3 and max=21. A higher value indicates greater influence over a partner.
Time Frame: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 51 | 59
score on a scale
  At 12 months | 17.1 (0.52) | 16.6 (0.51)
  Baseline / Pre-Intervention | 16.0 (0.56) | 15.0 (0.66)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.50, count GEE

14. Secondary Outcome: Empowerment: Personal
Description: Empowerment Scale: Personal. The theoretical minimum and maximum values are min=3 and max=21. A higher value indicates greater personal empowerment.
Time Frame: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 51 | 59
score on a scale
  At 12 months | 18.2 (0.40) | 18.3 (0.46)
  Baseline / Pre-Intervention | 18.6 (0.44) | 18.3 (0.46)

15. Secondary Outcome: Sexual Assertiveness: Refusal
Description: Sexual Assertiveness Refusal subscale. The theoretical minimum and maximum scores are min=6 and max=30. Higher scores indicate greater assertiveness in refusing sexual activity (better outcome).
Time Frame: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 51 | 59
score on a scale
  Baseline / Pre-Interveniton | 23.2 (0.87) | 24.4 (0.70)
  At 12 months | 25.0 (0.98) | 25.3 (0.77)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.86, count GEE

16. Secondary Outcome: Sexual Assertiveness: Prevent
Description: Sexual Assertiveness Prevent subscale. The theoretical minimum and maximum scores are min=6 and max=30. Higher scores indicate greater assertiveness in taking measures to prevent pregnancy (better outcome).
Time Frame: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 51 | 59
score on a scale
  Baseline / Pre-Intervention | 26.8 (0.68) | 25.8 (0.68)
  At 12 months | 27.1 (0.71) | 26.4 (0.59)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.46, count GEE

17. Other Pre Specified Outcome: Mother Adolescent Communication: Open Family Communication (Mother)
Description: Mother Adolescent Communication: Open Family Communication (Mother). The theoretical minimum and maximum values are min=10 and max=50. A higher value indicates greater mother-adolescent open family communication which is a better outcome.
Time Frame: 12 months
Population: Analyses were performed after multiple imputation for missing data. Number at 12 months before imputation were n=48 mothers for Risky sex prevention and n=54 mothers for Health behaviors.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 48 | 54
score on a scale
  Baseline / Pre-Interveniton | 41.4 (0.80) | 41.2 (0.76)
  At 12 months | 41.0 (0.93) | 41.5 (0.80)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.70, linear GEE

18. Other Pre Specified Outcome: Maternal Monitoring Scale (Mother)
Description: Maternal Monitoring Scale (Mother). The theoretical minimum and maximum values are min=8 and max=40. A higher value indicates greater maternal monitoring which is a better outcome.
Time Frame: 12 months
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 48 | 54
score on a scale
  Baseline / Pre-Interveniton | 37.1 (0.44) | 37.3 (0.35)
  At 12 months | 37.9 (0.29) | 37.4 (0.39)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.29, linear GEE

19. Other Pre Specified Outcome: Communication About Sex Self-Efficacy Scale
Description: Communication about Sex Self-Efficacy Scale. The theoretical minimum and maximum scores are min=12 and max=60. Higher scores indicate greater self-efficacy (better outcome).
Time Frame: 12 months
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risky Sex Prevention | Healthy Behaviors
Number analyzed (Participants) | 48 | 54
score on a scale
  Baseline / Pre-Interveniton | 56.0 (0.74) | 55.5 (0.92)
  At 12 months | 57.8 (0.59) | 58.3 (0.31)
Statistical Analysis 1: Comparison: Risky Sex Prevention vs Healthy Behaviors; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.43, linear GEE

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Risky Sex Prevention-Daughters: education, activities, empowerment, racial pride building
  Education, activities, empowerment, racial pride building: Intervention focuses on information aimed toward reducing or preventing risky sex behaviors of minority adolescent females.
- Healthy Behaviors-Daughters: General health education, activities
  General Health education, activities: Intervention focuses on information regarding general health knowledge and healthy behaviors (not including sex).
- Risky Sex Prevention-Mothers: Activities, empowerment
Arm/Group | Risky Sex Prevention-Daughters | Healthy Behaviors-Daughters | Risky Sex Prevention-Mothers | Healthy Behaviors-Mothers
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/59 | 0/48 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/59 | 0/48 | 0/54
Other Adverse Events (participants affected / at risk) | 0/51 | 0/59 | 0/48 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT02103218/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT02103218/SAP_001.pdf